CLINICAL TRIAL: NCT06326359
Title: Evaluation of Safety and Efficacy of Autologous Stromal Vascular Fraction Derived From Denovo Versus Platelet Rich Plasma Enhanced Donner Site in Treatment of Male Androgenic Alopecia
Brief Title: Autologous Stromal Vascular Fraction in Treatment of Male Androgenic Alopecia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Dina Ahmed Mahmoud, assistant lecturer, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Soh-Med-24-02-03MD
Record Dates: First submitted 2024-03-09; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Androgenic Alopecia
Keywords: autologous stromal vascular fraction; platelet rich plasma; male androgenic alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- autologous stromal vascular fraction derived from denovo (Active Comparator): autologous stromal vascular fraction derived from denovo in male androgenic alopecia
  Interventions: Procedure: autologous stromal vascular fraction
- autologous stromal vascular fraction after platelet rich plasma enhanced donner site (Active Comparator): autologous stromal vascular fraction after platelet rich plasma enhanced donner site in male androgenic alopecia
  Interventions: Procedure: autologous stromal vascular fraction

INTERVENTIONS:
Procedure: autologous stromal vascular fraction — autologous stromal vascular fraction injection as 2 sessions with 1 month interval at arm 1 arm 2: will receive 2 sessions of PRP with 3 weeks interval followed by stromal vascular fraction injection as 2 sessions with 1 month interval

SUMMARY:
Evaluation of Safety and efficacy of autologous stromal vascular fraction derived from denovo versus platelet rich plasma enhanced donner site in treatment of male androgenic alopecia

DETAILED DESCRIPTION:
40 Patients with androgenic alopecia will be randomly divided into 2 groups Group A (20): will receive 2 session of stromal vascular fraction directly after fat harvesting and processing and stromal vascular fraction extraction with 1 month interval .

Group B(20): will be injected with 2 session of Platelet rich plasma 3weeks interval at site of fat harvesting and will be followed 1 month later with fat aspiration from site where Platelet rich plasma was previously injected and this fat will undergo fat processing and stromal vascular fraction extraction followed by 2 session of stromal vascular fraction injection at scalp 1month interval .

Patients at both groups will receive topical and systemic antibiotics after stromal vascular fraction injection .

ELIGIBILITY:
Inclusion Criteria:

* Male patients with androgenic alopecia

Exclusion Criteria:

* Patients with other hair loss disorders as telogen effluvium, anagen effluvium, alopecia areata, cicatricial alopecia and trichotillomania.

Any other cutaneous disease as patients suffering from dermatological condition or a significant scarring in the treatment area.

Any systemic disease as autoimmune disorders , cardiac hepatic and renal patients.

patients who received minoxidil or any other oral, topical medications (including herbal medications) or injection procedures for the treatment of hair loss within 6 months prior to the study, or finasteride or dutasteride within 12 months of the study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
hair density | at baseline and at 6 month after treatment
  Trichoscopy
hair shaft thickness | at baseline and at 6 month after treatment
  TrichoScan

IPD SHARING:
Plan to Share IPD: No